CLINICAL TRIAL: NCT01126593
Title: Efficacy of Continuous Subacromial Bupivacaine Infusion for Postoperative Analgesia After Arthroscopic Rotator Cuff Repair.
Brief Title: Post-Op Rotator Cuff Pain Study With Subacromial Bupivacaine Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Principal Investigator, Paula J. Harriott, Orthopedic surgeon, Orlando Orthopaedic Center, Orlando Health, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 708009
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Bupivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo group (Placebo Comparator): The placebo group will receive the same subacromial infusion catheter as the study group.However, the reservoir will be filled with 200cc of 0.9% normal saline.
  Interventions: Drug: Normal Saline
- Control group (No Intervention): The control group patients will receive no continuous infusion catheter.
- Study Group (Experimental): Study group patients will receive a subacromial continuous standard spring loaded infusion catheter with 200cc of 0.5% bupivacaine in its reservoir. The infusion rate will be 4cc per hour.
  Interventions: Drug: 0.5% bupivacaine

INTERVENTIONS:
Drug: 0.5% bupivacaine — Study group patients will receive a subacromial continuous standard spring loaded infusion catheter with 200cc of 0.5% bupivacaine in its reservoir. The bupivacaine will have an infusion rate of 4cc an hour.
  Other Names: Marcaine
  Arms: Study Group
Drug: Normal Saline — The placebo group will receive the same subacromial infusion catheter however, the reservoir will be filled with 200cc of 0.9% Normal Saline.
  Other Names: Saline
  Arms: Placebo group

SUMMARY:
Subacromial pain catheters have been used with uncertain efficacy for many years after rotator cuff repair to aid in postoperative pain control. Our null hypothesis is that postoperative subacromial continuous infusion bupivacaine catheters will provide no pain control benefits over placebo infusions or no catheter use.

DETAILED DESCRIPTION:
This will be a prospective, randomized, double-blinded placebo controlled study. Randomization will be performed by a random numbers table. Envelopes will be sealed with the accompanying randomization group.Patients will be eligible for inclusion in the study if they have a full-thickness rotator cuff tear that has been deemed reparable by preoperative MRI. They will be included in the study if they are medically stable to undergo the surgery and consent to involvement in the study.

Patients consenting to the study will undergo arthroscopic rotator cuff repair by one of the two senior authors. The surgery will be performed as an outpatient procedure under general anesthesia. The procedure will be performed utilizing the standard techniques of the senior authors. All concomitant pathology found at the time of arthroscopy will be treated in the usual appropriate fashion. At the completion of the rotator cuff repair, patients will be randomly allocated to one of three groups. This will be done by opening a sealed envelope with the randomization allocation. The patients will either be placed into the study group, the placebo group or the control group.

ELIGIBILITY:
Inclusion Criteria:

* Full thickness rotator cuff tear
* Pre operative MRI
* Patients who are medically stable to undergo the surgery
* Patients who consent to involvement in the study

Exclusion Criteria:

* Prior surgery on the involved shoulder
* Preoperative MRI suggesting that the rotator cuff tear is unrepairable
* Patients with known allergies to oxycodone, bupivacaine or a similar drug
* Workman's compensation patients
* Patients who do not fill out their visual analog scores or their medication diaries.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Schwartzberg, MD, Principal Investigator — Orlando Orthopaedic Center and Orlando Health, Inc.
Locations (1):
- Orlando Orthopaedic Center, Orlando, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Principal investigator recruited patients in clinic.
Pre-assignment Details: If patient met the inclusion criteria and agreed to participate, they were given the consent to sign and were randomized into the trial.
Period: Overall Study
Arm/Group | Placebo Group | Control Group | Study Group
Started | 33 | 29 | 34
Completed | 29 | 27 | 32
Not Completed | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Control Group | Study Group | Total
Number analyzed (Participants) | 29 | 27 | 32 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (0.9) | 58 (0.6) | 56 (0.8) | 57 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 15 | 33
  Male | 20 | 18 | 17 | 55
Region of Enrollment [Number; unit: participants]
  United States | 29 | 27 | 32 | 88

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores
Description: Pain was measured via Visual Analong Scale in measurement (0-100mm).
Time Frame: O hour, 1, 2, 3, 4, 5, 6, 12 and 72 hours.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Group | Control Group | Study Group
Number analyzed (Participants) | 29 | 27 | 32
mm
  Pain at baseline | 64.7 (25.9) | 43.9 (33.6) | 51.4 (31.1)
  Pain at 1 hour | 60 (19.5) | 59.7 (26.5) | 52.3 (25.8)
  Pain at 2 hours | 60.5 (23.2) | 62 (26.0) | 50.7 (24.2)
  Pain at 3 hours | 60 (24.5) | 55.3 (27.1) | 51.2 (27.6)
  Pain at 4 hours | 52.6 (26.5) | 50.3 (28.7) | 46.8 (27.3)
  Pain at 5 hours | 54.5 (25.5) | 48.6 (24.1) | 46.7 (33.2)
  Pain at 6 hours | 42.9 (26.6) | 37.3 (22.3) | 42.2 (32.0)
  Pain at 12 hours | 46.6 (28.0) | 35.8 (22.7) | 42.8 (29.0)
  Pain at 72 hours | 45.0 (18.7) | 41.1 (18.1) | 42.7 (19.2)

ADVERSE EVENTS:
Time Frame: Adverse events were assesed for 6 months.
Arm/Group | Placebo Group | Control Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/29 | 0/34
Other Adverse Events (participants affected / at risk) | 0/33 | 0/29 | 0/34

LIMITATIONS AND CAVEATS:
It is possible that different catheter infusion rates, different bupivacaine concentrations, and pain modulation agents different from bupivacaine could result in different findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days